CLINICAL TRIAL: NCT04427670
Title: Implementation and Feasibility Study of Group Intervention for Individuals with Dysarthria Following Stroke and Their Carers in Pakistan
Brief Title: Group Intervention Study for Individuals with Dysarthria Following Stroke and Their Carers in Pakistan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isra University (Other)
Responsible Party: Principal Investigator, Saima maratab, principle investigator, Isra University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201/2020
Record Dates: First submitted 2020-03-14; First posted 2020-06-11 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Dysarthria As Late Effect of Stroke
Keywords: Stroke; Dysarthia; Intervention
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: RCT with intervention having experimental group. random Allocation of participants.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Regular speech therapy (Other): Regular speech therapy will be provided to the controlled group.
  Interventions: Other: Regular speech therapy
- Group intervention (Other): Group intervention will be provided to the experimental group.
  Interventions: Other: Group intervention

INTERVENTIONS:
Other: Group intervention — Group intervention programme designed for stroke survivors with dysarthria and their carers. The programme was eight weeks long, with weekly two sessions, each session lasting for two hours, lead by speech language therapist and was comprised of activities which addressed participants education about their dysarthria and stroke. The role of family , peer and professional was to provide support and communication practice.
  Arms: Group intervention
Other: Regular speech therapy — Regular speech therapy will be provided to the controlled group.Regular speech therapy is one to one speech therapy session,conducted twice a week for the duration of eight weeks.This intervention is implemented to patients with dysarthria following stroke in a format of one patient and one therapist per session.
  Arms: Regular speech therapy

SUMMARY:
Dysarthria is a common problem in Pakistan. therefore the current study aims to translate the dysarthria communication tools into urdu language for better understanding the population and the problem

DETAILED DESCRIPTION:
Dysarthria is the inefficiency or restricted capability to form intelligible speech because of the inability of motor control on the speech structures. There are many therapeutic approaches in Pakistan that are in use for the patients with dysarthria following stroke. One of them is one to one intervention which may include one dysarthria client along with the speech therapist. The therapist delivers step by step instructions to the client. The essential assessments are being held to initiate the treatment. The application of this intervention approach leaves some drawbacks, such as, the patients find it difficult to relate and adapt to the treatment offered. Generalization also seems to be complicated. The patients express a lack in motivation and support. The other mode of approach is group intervention, in which multiple dysarthria clients along with their caregivers & speech therapist are included. In the later one, there are greater chances of recovery for patients as they get peer support and build confidence through newfound friends, peer communication with realistic social setting, learning through teaching, increased awareness of skills and it is time constraints. The culture of practicing group sessions with dysarthria patients is lacked in Pakistan, which intends to meet and compensate for all the drawbacks and lacks of one on one intervention. By including the Dysarthria patients, therapist and the caregivers in the group intervention, there're greater chances of reduced anxiety for both patients & caregivers regarding disorder & its recovery.

ELIGIBILITY:
Inclusion Criteria:

1. 40 to 70 years age ranges
2. History of dysarthria previous six monthes
3. Primary level of education
4. Functional hearing and visual ablities -

Exclusion Criteria:

1. Patient with age below 40 to 70
2. Patients with diagnosis severe psychological illness
3. Patient with developmental dysarthria
4. Patient who come alone without any attendent

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2024-07-12 (Actual)

PRIMARY OUTCOMES:
efficacy of group intervention for Patients With Dysarthria will be assessed by the translated version of Roberston Dysarthria Profile. | 6 months
  Roberston Dysarthria Profile take responses on 5 point likert scale where 1 for worst and 5 for better outcome.
efficacy of group intervention for Patients With Dysarthria will be assessed by translated version of Communication Effectivness Measure | 6 months
  Communication Effectivness Measure is seven point scale arranging from 1 to 7 where 1 for worst outcome and 7 for better outcome.
Efficacy of group intervention for Patients With Dysarthria will be assessed by the translated version of Communicative Participation Item Bank. | 6 months
  Communicative Participation Item Bank is four point scale arranging from 0 to 3 where 0 for better communication participation and 3 for worst communication participation.
Efficacy of group intervention for Patients With Dysarthria will be assessed by Gernal Health Questionnaire | 6 months
  Gernal Health Questionnaire is four point scale in which responses 1 means better and 4 for worst condition
Efficacy of group intervention for Patients With Dysarthria will be assessed by Speech Intelligiblity Test | 6 months
  Speech Intelligiblity Test is three point scale where 2 stands for correct utterances and 0 shows wrong production of sounds.

CONTACTS AND LOCATIONS:
Overall Officials: Saima M Ali, PhD, Principal Investigator — Isra University, Islamabad
Locations (1):
- Sheikh Zayed medical Complex, Lahore, Punjab Province, Pakistan